CLINICAL TRIAL: NCT01106027
Title: A Single Center, Open-label Study to Determine the Safety and Efficacy of a Dosing Regimen of Eculizumab Added to Conventional Treatment in the Prevention of Acute Humoral Rejection (AHR) in Positive Crossmatch Deceased Donor Kidney Transplantation
Brief Title: Dosing Regimen of Eculizumab Added to Conventional Treatment in Positive Crossmatch Deceased Donor Kidney Transplant
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Difficulty enrolling; competing industry-funded multi-center clinical trial
Sponsor: Mayo Clinic (Other)
Collaborators: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Mark Stegall, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 09-005627DD
Record Dates: First submitted 2010-03-29; First posted 2010-04-19 (Estimated); Results first posted 2017-11-14 (Actual); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Kidney Transplant
MeSH Terms: interventions — eculizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Eculizumab (Experimental): Patients will be given 1200 mg of eculizumab intravenously over 30 minutes, 1 hour prior to surgery. Patients will be given 900 mg of eculizumab on Day 1 post-transplant. Patients will then be given 900 mg of eculizumab weekly through 4 weeks post-transplant.
  At week 4, patients will be assessed for donor specific anti-donor human leukocyte antigen (HLA) antibody (DSA). Patients with total DSA normalized values <5000 will stop eculizumab treatment. Patients with total DSA normalized values >5000 will continue eculizumab treatment every 14 days from week 5 through week 9. The dose will be increased to 1200 mg and dosing will now be every 2 weeks instead of weekly.
  Interventions: Drug: Eculizumab

INTERVENTIONS:
Drug: Eculizumab — Eculizumab 900 mg and 1200 mg, administered intravenously (IV)
  Other Names: Soliris

SUMMARY:
The purpose of this study is to test whether a dosing regimen of eculizumab in addition to standard posttransplant care in positive crossmatch deceased donor kidney transplant recipients will reduce the incidence of acute humoral rejection (AHR).

Patients included in this study will be those who have demonstrable anti-human leukocyte antigen (HLA) antibody specific for their deceased donor. It is our hypothesis that blockade of terminal complement activation with eculizumab at the time of transplant in combination with our current protocols will reduce the incidence of AHR in recipients of deceased donor kidney transplants who have anti-donor HLA antibody

DETAILED DESCRIPTION:
A strongly positive crossmatch has long been considered an absolute contraindication to kidney transplantation and most patients with anti-HLA antibody never were able to receive a kidney transplant. Over the past decade, significant progress has been made in overcoming early antibody-mediated renal allograft injury. Despite our best efforts, transplantation in these patients is still complicated by a high rate of acute humoral rejection.

While we have successfully transplanted more than 250 patients with DSA using living donors, applying these protocols to recipients of deceased donors has been problematic. This primarily is due to the fact that in contrast to living donation, the timing of a deceased donor kidney transplant cannot be planned. This leads to inadequate time to perform the multiple pretransplant plasmapheresis treatments needed to achieve a safe level of DSA at transplant. Thus, there is a major unmet need to develop therapy that will allow for the successful transplantation of deceased donor kidneys in recipients who have DSA.

* At the time of deceased donor kidney transplantation, patients will undergo one plasmapheresis prior to surgery.
* Patients will be given 1200 mg of eculizumab intravenously over 30 minutes, 1 hour prior to surgery.
* Patients will be given 900 mg of eculizumab on Day 1 post-transplant.
* Patients will then be given 900 mg of eculizumab weekly through 4 weeks post-transplant
* At week 4, patients will be assessed for DSA. Patients with total DSA normalized values <5000 will stop eculizumab treatment. Patients with total DSA normalized values >5000 will continue eculizumab treatment every 14 days from week 5 through week 9. The dose will be increased to 1200 mg and dosing will now be every 2 weeks instead of weekly. Similar "discontinuation assessments" will be performed at week 9, 26, 39 and 52.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* Has end stage renal disease (ESRD) and is to receive a kidney transplant from a deceased donor (DD) to whom he/she has a positive T or B cell crossmatch >200 at the time of transplant and DSA demonstrated by solid phase assays.
* Willing to comply with the protocol
* Females of child-bearing potential must have a negative pregnancy test (serum β-HCG) and sexually active females must agree to use a reliable and medically approved method of contraception
* Willing and able to give written informed consent
* Vaccinated against Neisseria meningitides (quadrivalent vaccine), Pneumococcus and H. influenzae at least two weeks prior to beginning desensitization

Exclusion Criteria:

* Unstable cardiovascular condition
* Previous splenectomy
* Active bacterial or other infection which is clinically significant in the opinion of the investigator
* Known or suspected hereditary complement deficiency
* Participation in any other investigational drug study or was exposed to an investigational drug or device within 30 days of randomization
* Pregnant, breast-feeding, or intending to conceive during the course of the study, including a one month follow-up period after drug discontinuation
* Known hypersensitivity to the treatment drug or any of its excipients
* History of illicit drug use or alcohol abuse within the previous year
* History of meningococcal disease
* Medical condition that, in the opinion of the investigator, might interfere with the patient's participation in the study, pose an added risk for the patient, or confound the assessment of the patient (e.g. severe cardiovascular or pulmonary disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-03 (Actual); Primary Completion 2016-08-19 (Actual); Study Completion 2016-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Stegall, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from Mayo Clinic in Rochester, Minnesota.
Period: Overall Study
Arm/Group | Eculizumab
Started | 2
Completed | 1
Not Completed | 1
Not completed — Lost graft early, discontinued | 1

BASELINE CHARACTERISTICS:
Arm/Group | Eculizumab
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Acute Humoral Rejection (AHR) up to One Year Post Transplant.
Description: Diagnosis of AHR will be based histological findings using Banff '05 criteria.
Time Frame: 1 year posttransplant
Population: The one subject who completed the study did not have acute humoral rejection. The other subject had the transplant but lost the graft early, meeting one of the endpoints of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 1
Participants | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Eculizumab
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eculizumab (N=2)
Acute antibody mediated rejection (Immune system disorders) | 1 (1)
Allograft nephrectomy (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eculizumab (N=2)
Presyncope (Cardiac disorders) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Peripheral edema (Cardiac disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated early due to difficulty enrolling and competing industry-funded multi-center clinical trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes